CLINICAL TRIAL: NCT06099704
Title: A Prospective, Observational Study of Canadian Patients Receiving Dupixent® for Moderate to Severe Atopic Dermatitis
Brief Title: Observational Study of Canadian Patients (6 Years or Older) Receiving Dupixent® for Moderate to Severe Atopic Dermatitis
Acronym: CANDID
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17843; U1111-1288-8240 (Other: WHO)
Record Dates: First submitted 2023-10-10; First posted 2023-10-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with msAD: Canadian msAD participants (ages 6+) who receive Dupixent for msAD according to the Canadian-country specific prescribing information (in accordance with the Canadian Dupixent Product Monograph)

SUMMARY:
This is a prospective, 18-month observational study of adult, adolescent and pediatric Canadian participants with Atopic Dermatitis (AD) commonly known as Eczema, who receive treatment with Dupixent for moderate-to-severe AD (msAD) according to the Canadian-specific prescribing information (in accordance with the Canadian Dupixent Product Monograph). The study will be conducted in approximately 30 centers in Canada to assess participants of all ethnicities and races. At each participating site, all AD participants who receive an initial prescription for Dupixent will be invited to participate in this study, until the Canadian enrollment goal is achieved.

DETAILED DESCRIPTION:
The duration of the study for each participant will be of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 6 years or older at baseline visit (Canada has received the country's regulatory approval for use of Dupixent treating msAD for these ages).
* Participant is initiating dupilumab as part of routine clinical care through the Dupixent Patient Support Program (PSP) for the treatment of msAD, as per reimbursement criteria. Decision to treat with dupilumab must have been reached prior to and independently of recruitment in the study.
* Have a physician's diagnosis of msAD.
* Provided signed informed consent or parental/legally acceptable representative consent and/or participant assent. During the study, subjects will continue to receive maintenance therapies for their AD as clinically indicated and as per usual medical practice.
* Participant or Parental representative able to understand English and/or Canadian French to complete study-related questionnaires.

Exclusion Criteria:

* Participants who have a contraindication to the drug according to the Canadian-specific prescribing information label.
* Any condition that, in the opinion of the Investigator, may interfere with participant's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other comorbidities that can predictably prevent the participant from adequately completing the schedule of visits and assessments.
* Participants currently participating in any interventional clinical trial which modifies participant care.
* Prior use of Dupixent within 6 months of the baseline visit.
* Participants not willing to sign the Informed Consent Form.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Canadian msAD participants (ages 6+) who receive Dupixent for msAD according to the Canadian-country specific prescribing information (in accordance with the Canadian Dupixent Product Monograph)
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving a reduction in Eczema Area and Severity Index (EASI) of at least 75% at 6 months | Month 6
  EASI is a validated measure used to assess the severity and extent of AD. Four AD disease characteristics [erythema, thickness (induration, papulation, and edema), scratching (excoriation), and lichenification] will each be assessed for severity by the Investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage of each body area assessed: head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0 (0%), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Total score is the sum of all subscores. EASI is a composite index with scores ranging from 0 to 72. Higher scores indicates worse condition. Data will be assessed to understand real-world effectiveness of Dupixent in a heterogeneic population of Canadian participants who initiate treatment for msAD using EASI score.
Percentage of participants achieving a reduction in EASI of at least 75% at 12 months | Month 12
  EASI is a validated measure used to assess the severity and extent of AD. Four AD disease characteristics [erythema, thickness (induration, papulation, and edema), scratching (excoriation), and lichenification] will each be assessed for severity by the Investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage of each body area assessed: head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0 (0%), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Total score is the sum of all subscores. EASI is a composite index with scores ranging from 0 to 72. Higher scores indicates worse condition. Data will be assessed to understand real-world effectiveness of Dupixent in a heterogeneic population of Canadian participants who initiate treatment for msAD using EASI score.
Percentage of participants achieving a reduction in EASI of at least 75% at 18 months | Month 18
  EASI is a validated measure used to assess the severity and extent of AD. Four AD disease characteristics [erythema, thickness (induration, papulation, and edema), scratching (excoriation), and lichenification] will each be assessed for severity by the Investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage of each body area assessed: head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0 (0%), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Total score is the sum of all subscores. EASI is a composite index with scores ranging from 0 to 72. Higher scores indicates worse condition. Data will be assessed to understand real-world effectiveness of Dupixent in a heterogeneic population of Canadian participants who initiate treatment for msAD using EASI score.

SECONDARY OUTCOMES:
Change from baseline in EASI score | From baseline to 6 months, 12 months, and 18 months post- Dupixent initiation
  Four AD disease characteristics [erythema, thickness (induration, papulation, and edema), scratching (excoriation), and lichenification] will each be assessed for severity by the Investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage of each body area assessed: head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0 (0%), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Total score is the sum of all subscores. EASI is a composite index with scoresEASI is a composite index with scores ranging from 0-72. Higher scores indicate worse conditions. Data will be assessed to understand (1) the real-world effectiveness of of Dupixent in a heterogeneic population and (2) to characterize disease burden and unmet need in Canadian participants who initiate treatment for msAD.
Change from baseline in Body Surface Area of Atopic Dermatitis Involvement (BSA) score | From baseline to 6 months, 12 months, and 18 months post- Dupixent initiation
  BSA affected by AD disease will be assessed for each major section of the body (head, neck, anterior trunk, back, upper limbs, lower limbs, and genitals). It will be reported as a percentage of all major body sections combined. Data will be assessed to understand (1) the real-world effectiveness of of Dupixent in a heterogeneic population and (2) to characterize disease burden and unmet need in Canadian participants who initiate treatment for msAD.
Change from baseline in Hospital Anxiety and Depression Scale (HADS) score | From baseline to 6 months, 12 months, 18 months post-Dupixent initiation
  HADS is a 14-item scale, with 7 items relating to anxiety and 7 relating to depression. Each item on the questionnaire is scored from 0-3. The anxiety/depression score is the sum of the scores of the 7 related items; one can score between 0 and 21 for either anxiety or depression. The total score is the sum of the scores of the 14 items ranging from 0 (no symptoms) to 42 (severe symptoms), with higher scores indicating higher nxiety/depression complains. Data will be assessed to understand (1) the real-world effectiveness of of Dupixent in a heterogeneic population and (2) to characterize disease burden and unmet need in Canadian participants who initiate treatment for msAD.
Change from baseline in Skin pain/soreness numerical rating scale (NRS) | From baseline to 6 months, 12 months, 18 months post-Dupixent initiation
  Skin pain NRS is a simple assessment tool asking participants to rate their skin pain or soreness using a 0 (No pain or soreness) to 10 (worst possible pain or soreness) NRS. Data will be assessed to understand (1) the real-world effectiveness of of Dupixent in a heterogeneic population and (2) to characterize disease burden and unmet need in Canadian participants who initiate treatment for msAD.
Change from baseline in skin feeling hot or burning NRS | From baseline to 6 months, 12 months, 18 months post-Dupixent initiation
  Skin burning NRS is a simple assessment tool asking participants to rate the sensation of their skin feeling hot or burning sensation using a 0 (Not feeling hot at all) to 10 (feeling extremely hot) NRS. Data will be assessed to understand (1) the real-world effectiveness of of Dupixent in a heterogeneic population and (2) to characterize disease burden and unmet need in Canadian participants who initiate treatment for msAD.
Change from baseline in Peak Pruritus NRS (PP-NRS) | From baseline to 6 months, 12 months, 18 months post-Dupixent initiation
  The peak pruritus NRS is a simple assessment tool asking participants to rate the intensity of their pruritis (itch) using a 0 (no itch) to 10 (worst possible itch) NRS. Data will be assessed to understand (1) the real-world effectiveness of of Dupixent in a heterogeneic population and (2) to characterize disease burden and unmet need in Canadian participants who initiate treatment for msAD.
Percentage of participants with Adverse Events (AEs) or Serious Adverse Events (SAEs) | From baseline up to 18 months post-Dupixent initiation
Reasons for discontinuation of Dupixent therapy | From baseline up to 18 months post-Dupixent initiation
  Data will be assessed to understand the real-world safety of Dupixent in a heterogeneic population of Canadian participants who initiate treatment for msAD
Mean time to Dupixent discontinuation | From baseline up to 18 months post-Dupixent initiation
  Data will be assessed to understand the real-world safety of Dupixent in a heterogeneic population of Canadian participants who initiate treatment for msAD
Median time to Dupixent discontinuation | From baseline up to 18 months post-Dupixent initiation
  Data will be assessed to understand the real-world safety of Dupixent in a heterogeneic population of Canadian participants who initiate treatment for msAD
Percentage of participants who initiated Dupixent and remained on treatment | At 3 months, 6 months, 12 months and 18 months post- Dupixent initiation
  Data will be assessed to understand the real-world safety of Dupixent in a heterogeneic population of Canadian participants who initiate treatment for msAD
Disease characteristics at baseline: EASI score | At baseline
  EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent. Four AD disease characteristics - erythema, thickness (induration, papulation, and edema), scratching (excoriation), and lichenification - will each be assessed for severity by the Investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage of each body area assessed: head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0 (0%), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Total score is the sum of all subscores. EASI is a composite index with scores. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Disease characteristics at baseline: BSA score | At baseline
  BSA affected by AD disease will be assessed for each major section of the body (head, neck, anterior trunk, back, upper limbs, lower limbs, and genitals). It will be reported as a percentage of all major body sections combined. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Disease characteristics at baseline: Time between diagnosis and Dupixent prescription | At baseline
  Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Change from baseline in sleep Disturbance NRS scores post-Dupixent initiation | From baseline to 3 months, 6 months, 12 months and 18 months post- Dupixent initiation
  Participants will be asked to report the severity of their sleep disturbance during the past 7 days using a 0 (sleep not disturbed at all) to 10 (sleep extremely disturbed) NRS. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Change from baseline in the dermatology life quality index (DLQI)/the Children's Dermatology Life Quality Index (CDLQI) scores post-Dupixent initiation | From baseline to 3 months, 6 months, 12 months and 18 months post- Dupixent initiation
  The DLQI and CDLQI are a 10-item validated questionnaire to assess the impact of AD disease on quality of life (QoL) in adults and adolescents/pediatrics, respectively. The rating scale range from 0 (not at all) to 3 (very much) 10 items, which assess QoL over the past week. The total score is the sum of all 10-items ranging from 0 to 30; a high score is indicative of a poor QoL. The CDLQI will be used for adolescent participants (aged ≥ 12 to < 18 years) and pediatric participants (aged ≥ 6 to < 12 years); these participants will switch to the DLQI when they turn 18 years of age (if this happens during the study). The CDLQI will be completed with help from participant's caregivers. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Change from baseline in Work Productivity and Activity Impairment Questionnaire for AD (WPAI-AD) scores post-Dupixent initiation | From baseline to 3 months, 6 months, 12 months and 18 months post- Dupixent initiation
  WPAI-AD is designed to assess the impact of AD disease on the participant's productivity. It is a 6-item validated questionnaire to measure effect of your AD disease on your ability to work and perform regular activities over a 7-day recall period. The questionnaire ask participants to recall following types of activities during the previous 7 days: absenteeism (time missed), presenteeism (impairment/ reduced effectiveness), productivity, and activity impairment. Total WPAI-AD outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. Caregivers complete the questionnaire for affected children. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Change from baseline in Work Productivity and Activity Impairment Questionnaire+Classroom Impairment Questions for AD (WPAI-CIQ-AD) scores post-Dupixent initiation | From baseline to 3 months, 6 months, 12 months and 18 months post- Dupixent initiation
  WPAI-CIQ-AD is designed to asses the impact of AD disease on the participant's productivity. It is a 9-item validated questionnaire to measure participants ability to work, attend classes, and perform regular daily activities during the previous 7 days. Participants are asked to report the work time or classes lost due to AD disease; the impact of eczema on the performance in the workplace, at school, or during university classes; the effect of eczema on other daily activities during the previous 7 days. Total WPAI-AD outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. Caregivers complete the questionnaire for affected children. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Change from baseline in Dermatitis Family Impact (DFI) score post-Dupixent initiation | From baseline to 3 months, 6 months, 12 months and 18 months post- Dupixent initiation
  DFI is a 10-question disease-specific measure to assess the impact of AD disease on the QoL of the parents and family members of affected children (≥ 6 to < 18 years)'. The DFI is calculated by summing the score of each question with a maximum total score of 30 (higher scores indicate higher impact on life of family). Caregivers complete the questionnaire for affected children. Data will be assessed to characterize disease burden and unmet need in Canadian msAD participants who initiate treatment with Dupixent.
Concomitant treatments received | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Dupixent dosing regimen | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Most commonly used Dupixent dosing regimens | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Dupixent treatment duration | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Number of gaps in Dupixent treatment | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Longest gap in Dupixent treatment | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Number of missed Dupixent doses over 18 months per participant | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
AD treatments to which participants switch when discontinuing dupixent | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Reasons for initiation of new AD treatments | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Reasons for discontinuation and/or switching AD treatments | From baseline up to 18 months
  Data will be assessed to describe real-world treatment patterns in Canadian msAD participants who initiate treatment with Dupixent
Change from baseline in HADS | From baseline to 6 months, 12 months and 18 months post- Dupixent initiation
  HADS is a 14-item scale, with 7 items relating to anxiety and 7 relating to depression. Each item on the questionnaire is scored from 0-3. The anxiety/depression score is the sum of the scores of the 7 related items; one can score between 0 and 21 for either anxiety or depression. The total score is the sum of the scores of the 14 items ranging from 0 (no symptoms) to 42 (severe symptoms), with higher scores indicating higher nxiety/depression complains. Data will be assessed to understand patterns and/or changes in non-atopic conditions in Canadian msAD participants who initiate treatment with Dupixen.
Change from baseline in sleep disturbance NRS scores post-Dupixent initiation | From baseline to 3 months, 6 months, 12 months and 18 months post- Dupixent initiation
  Participants will be asked to report the severity of their sleep disturbance during the past 7 days using a 0 (sleep not disturbed at all) to 10 (sleep extremely disturbed) NRS. Data will be assessed to understand patterns and/or changes in non-atopic conditions in Canadian msAD participants who initiate treatment with Dupixent.
Change from baseline in height | From baseline to 6 months, 12 months and 18 months post- Dupixent initiation
  Data will be assessed to understand patterns and/or changes in non-atopic conditions in Canadian msAD participants who initiate treatment with Dupixent
Change from baseline in weight | From baseline to 6 months, 12 months and 18 months post- Dupixent initiation
  Data will be assessed to understand patterns and/or changes in non-atopic conditions in Canadian msAD participants who initiate treatment with Dupixent
Change from baseline in BMI | From baseline to 6 months, 12 months and 18 months post- Dupixent initiation
  Data will be assessed to understand patterns and/or changes in non-atopic conditions in Canadian msAD participants who initiate treatment with Dupixent
Number of participants with demographic characteristics | From baseline up to 18 months
  Data will be assessed for all demographic characteristics by age, sex, race and ethnicity, location to understand baseline characteristics and/or changes in Canadian msAD participants who initiate treatment with Dupixent, with co-existing type 2 inflammatory diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (29):
- Canada (29):
  - Investigational Site Number : 1240019, Calgary, Alberta
  - Investigational Site Number : 1240021, Calgary, Alberta
  - Investigational Site Number : 1240009, Edmonton, Alberta
  - Investigational Site Number : 1240007, Edmonton, Alberta
  - Investigational Site Number : 1240028, Nanaimo, British Columbia
  - Investigational Site Number : 1240010, Surrey, British Columbia
  - Investigational Site Number : 1240029, Winnipeg, Manitoba
  - Investigational Site Number : 1240026, Fredericton, New Brunswick
  - Investigational Site Number : 1240020, Halifax, Nova Scotia
  - Investigational Site Number : 1240002, Ajax, Ontario
  - Investigational Site Number : 1240024, Barrie, Ontario
  - Investigational Site Number : 1240031, Cobourg, Ontario
  - Investigational Site Number : 1240011, Etobicoke, Ontario
  - Investigational Site Number : 1240016, London, Ontario
  - Investigational Site Number : 1240025, Newmarket, Ontario
  - Investigational Site Number : 1240008, Peterborough, Ontario
  - Investigational Site Number : 1240005, Richmond Hill, Ontario
  - Investigational Site Number : 1240033, Toronto, Ontario
  - Investigational Site Number : 1240030, Toronto, Ontario
  - Investigational Site Number : 1240014, Toronto, Ontario
  - Investigational Site Number : 1240018, Waterloo, Ontario
  - Investigational Site Number : 1240034, Whitby, Ontario
  - Investigational Site Number : 1240012, Montreal, Quebec
  - Investigational Site Number : 1240017, Montreal, Quebec
  - Investigational Site Number : 1240006, Pointe-Claire, Quebec
  - Investigational Site Number : 1240013, Québec, Quebec
  - Investigational Site Number : 1240023, Saint-Jean-sur-Richelieu, Quebec
  - Investigational Site Number : 1240003, Regina, Saskatchewan
  - Investigational Site Number : 1240027, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org